CLINICAL TRIAL: NCT05960201
Title: A Phase 2, Open-label, Non-randomized, Single-center Study to Explore the Diagnostic Performance of [18F]FES PET/CT for the Assessment of Axillary Lymph Node Metastasis in Invasive Lobular Carcinoma of the Breast
Brief Title: Diagnostic Performance of [18F]FES PET/CT for Axillary LN Metastasis in Invasive Lobular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sangwon Han, Clinical assistant professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FES lobular
Record Dates: First submitted 2023-07-18; First posted 2023-07-25 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Carcinoma, Lobular
MeSH Terms: conditions — Carcinoma, Lobular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- invasive lobular breast cancer (Experimental): images for 90 minutes after F-18 FES injection
  Interventions: Drug: [18F]fluoroestradiol (FES)

INTERVENTIONS:
Drug: [18F]fluoroestradiol (FES) — F-18 FES 111~222 MBq(megabecquerel) injection

SUMMARY:
This study aims to explore the diagnostic validity of [18F]FES PET/CT for the evaluation of axillary lymph node metastasis in patients with invasive lobular breast cancer having clinically suspected or confirmed axillary lymph node metastasis.

DETAILED DESCRIPTION:
Invasive lobular carcinoma (ILC) is known to account for about 10-15% of all invasive breast cancer and is the second most common subtype of breast cancer following invasive ductal carcinoma (IDC). ILC is histologically characterized by the loss of E-cadherin involved in cell adhesion, which contributes to the growth and infiltration of tumors in the characteristic non-adhesive single cell layer pattern of ILC]. Therefore, ILC often has no tumors detected by physical examinations and the sensitivity of mammography being reported to be 34%, which is much lower than IDC (81%). Therefore, the diagnosis of ILC is often delayed, the tumor size is larger and the stage is higher than that of IDC at the first visit. The diagnostic accuracy of breast ultrasound for axillary lymph node metastasis is reported as 55-92% for sensitivity and 80-97% for specificity. However, in the case of ILC, the diagnostic performance is significantly lower than this. According to the previous study on ILC, mammography had 7% of sensitivity, ultrasound had 26%, and MRI had 7% in diagnosing axillary lymph node metastasis with 38% of patients having false positive results for axillary lymph node metastasis. This is related to ILC-specific metastasis patterns in which only cells are replaced by cancer cells while maintaining the normal structure of the lymph node and the absence of desmoplastic reaction. The NCCN guideline recommends that during axillary lymph node resection, resection is performed up to level III if lymph node metastasis is confirmed or suspected in axillary level II or III. Preoperative chemotherapy should be considered for lymph node metastasis of cN3 or Bulky or matted cN2 stage. Considering the limited diagnostic accuracy of those standard imaging tests for diagnosis of axillary lymph node metastasis, [18F]FES PET/CT may help change treatment strategy, such as changing the extent of axillary lymph node resection or performing neoadjuvant chemotherapy instead of upfront surgery in patients with ILC. In addition, considering that high rate of distant metastasis and limited diagnostic accuracy of preexisting imaging modality in ILC, [18F]FES PET/CT is likely to help treatment decision making by discovering unexpected distant metastases. It is reported that the implementation of [18F]FES PET/CT contributed to the change in treatment policy in about 26% of patients compared to conventional standard imaging and [18F]FDG PET/CT. Currently in South Korea, reimbursement of [18F]FES PET/CT is limited to patients with recurrent or metastatic breast cancer whose lesions are located in the cervical spine, upper thoracic, pelvic, peritoneum, pleural, and mediastinal lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 19 years or older regardless of race/ethnicity.
* Subjects with histologically confirmed estrogen receptor-positive invasive lobular breast cancer within 90 days prior to [18F]FES PET/CT imaging
* Subjects whose primary tumor of cT1-3 according to the American Joint Committee on Cancer (AJCC) 8th tumor staging system
* Subjects with suspected or confirmed axillary lymph node metastasis clinically or in imaging test (ultrasound)
* Subjects who scheduled to undergo sentinel node biopsy or axillay lymph node dissection within 90 days of [18F]FES PET/CT imaging
* Subjects whose Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 2 points or less

Exclusion Criteria:

* Subject or the subject's legally acceptable representative does not provide written informed consent form
* Subjects with confirmed or suspected large, bulky, matted cN2 or cN3 axillary lymph node metastases, or distant metastases.
* Previous history of ipsilateral axillary lymph node dissection, sentinel lymph node surgery, or lymph node dissection biopsy.
* Patients who are scheduled for or have undergone chemotherapy, radiotherapy, antihormone therapy, targeted therapy, or immunotherapy between [18F]FES PET/CT and pathological diagnosis
* Subjects who are pregnant or lactating. Exclusion of the possibility of pregnancy is made by one of the following: 1) Physiologically menopausal (menstruation has stopped for more than 2 years), 2) Surgically infertility (with a history of bilateral oophorectomy or hysterectomy), 3) In the case of subjects with a possibility of pregnancy, negative serum or urine pregnancy test before administration of [18F]FES has to be negative within 24 hours, and the subjects are instructed to use contraception during her participation in this study.
* Subject has concurrent severe and/or uncontrolled and/or unstable medical condition other than cancer (e.g., congestive heart failure, acute myocardial infarction, severe lung disease, chronic kidney disease or chronic liver disease).
* Subject is a relative or student of the investigator or otherwise in a dependent relationship
* Subject has already participated in this study
* Subject not being able to provide intact data for this study due to personal circumstances or other reasons in the judgment of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Patient based sensitivity, specificity, positive predictive and negative predictive values of a qualitative [18F]FES PET/CT assessment of axillary lymph node metastasis | 90-120 min
  diagnostic accuracy of qualitative [18F]FES PET/CT analysis

SECONDARY OUTCOMES:
Patient based sensitivity, specificity, positive predictive and negative predictive values of quantitative [ 18 F]FES PET/CT evaluation for axillary lymph node metastasis | 90-120 min
  diagnostic accuracy of quatitative [18F]FES PET/CT analysis
Patient based sensitivity, specificity, positive predictive and negative predictive values of [18F]FES PET/CT in FNA or CNB-negative patients | 90-120 min
  Subgroup analsis of FNA or CNB-negative patients
Detection rate of qualitative [18F]FES PET/CT evaluation for cN3 lymph node metastasis | 90-120 min
  Unexpected N3 node detection rate
Detection rate of qualitative [18F]FES PET/CT evaluation for distant metastasis | 90-120 min
  Unexpected M1 detection rate

CONTACTS AND LOCATIONS:
Overall Officials: Sangwon Han, Principal Investigator — Clinical assistant professor
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No